CLINICAL TRIAL: NCT06291532
Title: Feasibility and Usability of a Virtual Reality System to Improve Standardized Rehabilitation in Patients With Moderate Intellectual Disability and Severe Autism Spectrum Disorder
Brief Title: Feasibility and Usability of a Virtual Reality System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesca Cucinotta, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRRS01
Record Dates: First submitted 2024-02-09; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (EG) (Experimental): The group consists of patients diagnosed with autism spectrum disorder and intellectual disability who underwent treatment with VRRS
  Interventions: Device: Rehabilitation with VRRS

INTERVENTIONS:
Device: Rehabilitation with VRRS — The patients underwent an experimental intervention lasting two months (9 sessions lasting about 40 minutes) integrated into the regular activity of a semi-residential center for autistic adolescents and young adults.
  The proposed exercises were 2D and the patient interacted with the scenarios through the touch screen. For all participants, the tasks were the same, but difficulty and duration varied according to the needs and goals to be achieved.

SUMMARY:
Intellectual disability (ID) and autism spectrum disorder (ASD) are often co-occurring neurodevelopmental disorders that require composite intervention. However, standardized rehabilitation programs presented several limitations due to behavioral problems and poor engagement in proposed activity. The Virtual Reality Rehabilitation System (VRRS) is a medical device is recognized as one of the most advanced systems to rehabilitate patients with motor, cognitive, linguistic and behavioral disorders. The use of VRRS offers the opportunity to adapting task parameters according to the patient's performance and the virtual system increases engagement and avoids boredom and frustration. the patients underwent a two months experimental intervention integrated into the regular activity of a semi-residential center for autistic adolescents and young adults.

ELIGIBILITY:
Inclusion criteria:

* subjects diagnosed with ASD and ID, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
* age between 6 and 40 years;
* cognitive level <65 Intellectual Quotient
* signed informed consent

Exclusion criteria:

* subjects without diagnosis of ASD and ID, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
* age not between 6 and 40 years;
* cognitive level >65 Intellectual Quotient
* unsigned informed consent

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Usability questionnaire | T0 (BASELINE) - T1 (SIX MONTHS)
  The questionnaire used a 5-point ordinal scale, where 5 is the most favorable score and 1 is the least favorable score; the score 3 corresponds to "no opinion". The questionnaire will be completed by all therapists at the end of the treatment.
Virtual Reality Rehabilitation System (VRRS) electromedical device parameters: screen attention time | T0 (BASELINE) -T1 (SIX MONTHS)
  During the execution of the exercise, the attention time maintained on the screen was recorded.
Virtual Reality Rehabilitation System (VRRS) electromedical device parameters: the number of repetitions of the exercises. | T0 (BASELINE) -T1 (SIX MONTHS)
  During the execution of the exercise, the number of repetitions of the exercises was recorded
Virtual Reality Rehabilitation System (VRRS) electromedical device parameters:global scores for exercise. | T0 (BASELINE) -T1 (SIX MONTHS)
  The total scores obtained were recorded during the execution of the exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy

REFERENCES:
- [Background] Bernard Paulais MA, Mazetto C, Thiebaut E, Nassif MC, Costa Coelho De Souza MT, Stefani AP, Blanc R, Gattegno MP, Aiad F, Sam N, Belal L, Fekih L, Kaye K, Contejean Y, Wendland J, Barthelemy C, Bonnet-Brilhault F, Adrien JL. Heterogeneities in Cognitive and Socio-Emotional Development in Children With Autism Spectrum Disorder and Severe Intellectual Disability as a Comorbidity. Front Psychiatry. 2019 Jul 19;10:508. doi: 10.3389/fpsyt.2019.00508. eCollection 2019. PMID 31396112
- [Background] De Luca R, Bonanno M, Rifici C, Pollicino P, Caminiti A, Morone G, Calabro RS. Does Non-Immersive Virtual Reality Improve Attention Processes in Severe Traumatic Brain Injury? Encouraging Data from a Pilot Study. Brain Sci. 2022 Sep 8;12(9):1211. doi: 10.3390/brainsci12091211. PMID 36138947